CLINICAL TRIAL: NCT04241146
Title: A Randomized Controlled Trial for Optimal Feeding Tube Placement
Brief Title: Optimal Feeding Tube Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Avanos Medical (Other)
Responsible Party: Principal Investigator, Andrew D. Meyer, Andrew Meyer, MD, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC20170704H
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Results first posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Enteral Feeding Intolerance
Keywords: enteral nutrition; radiation exposure; nursing care; pediatrics; radiation, non-ionizing
MeSH Terms: interventions — Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard Blind Technique of Tube placement (Active Comparator): FDA approved technique of enteral nutrition tube placement
  Interventions: Device: Enteric Tube
- CORTRAK enteral access system (CEAS) placement (Active Comparator): An electromagnetic device used to enable enteral nutrition tube placement
  Interventions: Device: CORTRAK enteral access system

INTERVENTIONS:
Device: Enteric Tube — A post pyloric feeding tube used in patients requiring enteral nutrition
  Other Names: Enteral nutrition tube
  Arms: Standard Blind Technique of Tube placement
Device: CORTRAK enteral access system — Electromagnetic guidance system for enteric feeding tube placement
  Other Names: CEAS
  Arms: CORTRAK enteral access system (CEAS) placement

SUMMARY:
A randomized controlled trial comparing current standard blind method to CORTRAK enteral access system (CEAS), an FDA approved electromagnetic device to place enteric tubes.

DETAILED DESCRIPTION:
Patient population would include patients in pediatric intensive care unit, pediatric cardiac unit, intermediate medical care unit and pediatric floor who receives postpyloric feeding tube placements. The study team are going to monitor total time and number attempts required for each successful placement, correlation of findings on x-ray versus CEAS, cost-effectiveness of this new equipment with standard blind method and decrease in radiation exposure with CEAS.

ELIGIBILITY:
Inclusion Criteria: Patient admitted to pediatric floor, intermediate care unit, pediatric intensive care unit, or congenital care unit requiring post-pyloric feeding tube placement of size eight french or more and not meeting any of exclusion criteria

Exclusion Criteria: Under three kilograms, Open chest wall, Open abdominal wall

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2018-01-06 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2019-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Meyer, MD, Principal Investigator — University of Texas Health San Antonio
Locations (1):
- University Hospital, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data is available to all researchers upon contact of sponsoring organization and investigator Andrew D. Meyer.
Supporting Information: Study Protocol
Time Frame: Data will be available after primary manuscript is accepted for publication.
Access Criteria: Data will be available in journal publication

REFERENCES:
- [Derived] Jha P, Rupp L, Bonilla L, Gelfond J, Shah JN, Meyer AD. Electromagnetic Versus Blind Guidance of a Postpyloric Feeding Tube in Critically Ill Children. Pediatrics. 2020 Oct;146(4):e20193773. doi: 10.1542/peds.2019-3773. PMID 32994178

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Blind Technique of Tube Placement | CORTRAK Enteral Access System (CEAS) Placement
Started | 24 | 28
Completed | 24 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects admitted to hospital requiring feeding tube placement
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Blind Technique of Tube Placement | CORTRAK Enteral Access System (CEAS) Placement | Total
Number analyzed (Participants) | 24 | 28 | 52
Age, Customized [Number; unit: participants]
  Age 0-1 years | 14 | 13 | 27
  Age 2-5 years | 4 | 9 | 13
  Age 6-10 years | 2 | 2 | 4
  Age 11-15 years | 1 | 0 | 1
  Age 16-18 years | 3 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 13 | 17 | 30
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 16 | 19 | 35
  White | 4 | 6 | 10
  Asian | 0 | 2 | 2
  Black, African American | 3 | 1 | 4
  Unknown | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 24 | 28 | 52

OUTCOME MEASURES:

1. Primary Outcome: Duration of Time
Description: Time taken for placement of enteral tube
Time Frame: Baseline to End of procedure up to 30 minutes
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Standard Blind Technique of Tube Placement | CORTRAK Enteral Access System (CEAS) Placement
Number analyzed (Participants) | 24 | 28
Minutes | 19 [9.25 to 27.0] | 2.5 [2.0 to 7.5]

2. Secondary Outcome: Number of X-Rays
Description: Number of X-rays required to achieve correct tube placement
Time Frame: Baseline to End of procedure up to 30 minutes
Measure: Mean (Full Range); unit: x-rays
Arm/Group | Standard Blind Technique of Tube Placement | CORTRAK Enteral Access System (CEAS) Placement
Number analyzed (Participants) | 24 | 28
x-rays | 2 [1 to 4] | 1 [1 to 1]

ADVERSE EVENTS:
Time Frame: Baseline to End of procedure (tube placement)
Arm/Group | Standard Blind Technique of Tube Placement | CORTRAK Enteral Access System (CEAS) Placement
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/28
Other Adverse Events (participants affected / at risk) | 0/24 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-21): https://cdn.clinicaltrials.gov/large-docs/46/NCT04241146/Prot_SAP_000.pdf